CLINICAL TRIAL: NCT03632044
Title: Evaluation of Trigeminal Nerve Blockade in the Pterygopalatine Fossa for Cleft Palate Repair: a Pilot Study
Brief Title: Evaluation of Trigeminal Nerve Blockade
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB201801011; OCR18511 (Other: University of Florida)
Record Dates: First submitted 2018-08-06; First posted 2018-08-15 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-11

CONDITIONS: Mouth Abnormalities; Cleft Palate; Birth Defect
MeSH Terms: conditions — Mouth Abnormalities; Cleft Palate; Congenital Abnormalities | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: This randomized, double-blinded study. Subjects will be randomly assigned to one of two different protocols by a designated study team member based on a computer generated randomization table. Randomization will occur following consent. Randomization will be 1:1.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: During the block placement the surgical team will be asked to leave the operating room briefly to remain blinded to the group assignment of all patients as the surgical team will manage the subjects post-operative care and determine discharge readiness.
  ICU nursing staff and parents will be informed of participation in the study but will not be informed as to group assignment to remain blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Suprazygomatic maxillary nerve blockade (Experimental): A single injection into the pterygopalatine fossa bilaterally of 0.2% ropivacaine at a dose of 0.15 mL/kg (block) after the induction of general anesthesia.
  Interventions: Drug: Ropivacaine
- 25 Gauge needle (Sham Comparator): Subcutaneous placement of a 25 Gauge needle as a sham comparator after the induction of general anesthesia. Nothing will be injected.
  Interventions: Other: Sham Comparator

INTERVENTIONS:
Drug: Ropivacaine — A single injection into the pterygopalatine fossa bilaterally of 0.2% ropivacaine at a dose of 0.15 mL/kg (block) after the induction of general anesthesia
  Other Names: Naropin
  Arms: Suprazygomatic maxillary nerve blockade
Other: Sham Comparator — The subcutaneous placement of a 25 Gauge needle as a sham control after the induction of general anesthesia. Nothing will be injected.
  Other Names: Control
  Arms: 25 Gauge needle

SUMMARY:
Cleft palate repair requires high doses of opioids for pain control postop. An alternative approach is placement of nerve blocks in the pterygopalatine fossa bilaterally, blocking the maxillary nerve & covering the entire midface. Application of bilateral suprazygomatic maxillary nerve blockade of the infraorbital nerve may provide effective analgesia for cleft lip repair, improving time to oral intake, pain control and time to hospital discharge.

DETAILED DESCRIPTION:
Cleft palate is a common congenital anomaly for which surgical repair is indicated during early childhood. The surgical repair of cleft palate is very painful, and generally requires high doses of opioids for adequate pain control, placing children at risk for post-operative respiratory depression and airway obstruction. An alternative approach to post-operative analgesia for cleft palate repair is the placement of nerve blocks in the pterygopalatine fossa bilaterally, blocking the maxillary nerve and covering the entire mid-face. This randomized, double-blinded study will investigate the utility of maxillary nerve blockade in controlling post-operative pain, decreasing opioid requirements, improving post-operative oral food and drink intake, and decreasing hospital length-of-stay after cleft palate repair.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting for palatoplasty for cleft palate only.
* Parent/guardian consents to participate
* Normal oral food and water intake before surgery
* No underlying chronic pain condition

Exclusion Criteria:

* Parent/guardian refuses to consent
* Patient requires revision surgery on the palate
* Patient requires surgery in addition to palatoplasty, including, but not limited to pharyngeal flap or soft palate lengthening procedures.
* Any underlying chronic pain condition
* Presence of any other factor which, at the discretion of any member of the study team, makes the patient a poor candidate for block placement.
* Presence of any other factor which, at the discretion of any member of the study team, makes the patient a poor candidate for research participation.
* History of Pierre Robin sequence
* Planned or anticipated need for any type of artificial airway post-op

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2018-11-20 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in time to oral intake following palatoplasty for cleft palate | Change from baseline (post-op) and through study completion, an average of 96 hours.
  Application of bilateral suprazygomatic maxillary nerve blockade of the infraorbital nerve to provide effective analgesia for cleft lip repair, improving time to oral intake after surgery.

SECONDARY OUTCOMES:
Change in amount of opioids following palatoplasty for cleft palate | Change from baseline (post-op) and through study completion, an average of 96 hours.
  Application of bilateral suprazygomatic maxillary nerve blockade of the infraorbital nerve to provide effective analgesia for cleft lip repair, improving pain control after surgery.
Change in length of hospitalization following palatoplasty for cleft palate | Change from baseline (post-op) and through study completion, an average of 96 hours.
  Application of bilateral suprazygomatic maxillary nerve blockade of the infraorbital nerve to provide effective analgesia for cleft lip repair, improving time to hospital discharge after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Cameron R Smith, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States